CLINICAL TRIAL: NCT01151761
Title: Phase II Study of Stereotactic Body Radiotherapy (SBRT) and Chemotherapy for Unresectable Cholangiocarcinoma Followed by Liver Transplantation
Brief Title: Phase II SBRT & Chemo for Unresectable Cholangiocarcinoma Followed by Liver Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel T. Chang, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP0032; HEP0032 (Other: Stanford University)
Record Dates: First submitted 2010-06-15; First posted 2010-06-28 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Cholangiocarcinoma; Hepatobiliary Neoplasm; Liver Cancer; Bile Duct Cancer; Cancer of Gallbladder
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Radiosurgery; Gemcitabine; Cisplatin; Carboplatin; Capecitabine; Fluorouracil; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT, Chemo and Liver Transplantation (Experimental): The patients received Stereotactic Body Radiotherapy and Chemotherapy followed by a liver transplantation. The chemo could be any combination of the following: Gemcitabine, Cisplatin, Carboplatin, Capecitabine and 5FU
  Interventions: Procedure: Stereotactic Body Radiotherapy; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Drug: Capecitabine; Drug: 5FU; Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Stereotactic Body Radiotherapy — Standard of care
  Other Names: External photon radiation
Drug: Gemcitabine — 100 mg/m2, IV
  Other Names: Gemzar
Drug: Cisplatin — 25 mg/m2, IV
  Other Names: Platinol; Platinol-AQ
Drug: Carboplatin — AUC 2, based on Calvert formula, IV
  Other Names: Paraplatin; Paraplatin-AQ
Drug: Capecitabine — 1000 mg/m2, PO
  Other Names: Xeloda
Drug: 5FU — 200 mg/m2
  Other Names: Fluorouracil; Adrucil; Carac; Efudix; Efudex; Fluoroplex
Procedure: Liver transplantation

SUMMARY:
The purpose of this study is to determine progression-free survival at 12 months for stereotactic body radiotherapy (SBRT) and chemotherapy for unresectable hilar cholangiocarcinoma (CCA).

DETAILED DESCRIPTION:
Investigators hope to learn more about neoadjuvant SBRT and chemotherapy for unresectable CCA, and if SBRT followed by chemotherapy can lead to successful liver transplantation. This knowledge is important for this patient group as this disease is a highly lethal malignancy that often presents as unresectable, however surgery or transplantation are the only curative options.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cholangiocarcinoma by any of the below:

  * Positive transcatheter biopsy or brush cytology
  * CA 19-9 ≥ 100mg/mL with a malignant-appearing stricture on cholangiography
  * Biliary ploidy by fluorescent in situ hybridization with a malignant stricture on cholangiography
* Liver tumors not to exceed 8 cm in greatest axial dimension (800 cc of uninvolved liver)
* Unresectable tumor above cystic duct
* Hepatic lesion in patients for whom surgical resection is not possible or would not result in an opportunity for cure by any of the below:

  * Bilateral segmental ductal extension
  * Encasement of the main portal vein
  * Unilateral segmental ductal extension with contralateral vascular encasement
  * Unilateral atrophy with either contralateral segmental ductal or vascular (hepatic artery, portal vein) involvement
* Ascites is allowed if the Model for End-Stage Liver Disease (MELD) score is <15[1]
* Age > 18 years old
* Eastern Clinical Oncology Group performance status 0, 1 or 2 (Appendix 1)
* Lab values within 2 wks prior to randomization:

  * See STUDY SCHEMA for specific blood count inclusion criteria: ANC ≥ 500 x 109/L (≥ 1500/mm3), Platelets ≥ 5 x 109/L (≥ 50,000/mm3), Hgb ≥ 9g/dL
  * Adequate liver function: Total bilirubin ≤1.5 x upper limit of normal (ULN); ALT and/or AST & alkaline phosphatase ≤ 5 x ULN.
  * Adequate biliary drainage, with no evidence of active uncontrolled infection (patients on antibiotics are eligible).
  * See STUDY SCHEMA for specific renal function inclusion criteria: Adequate renal function with a calculated GFR ≥ 40 ml/min. If the calculated GFR is below 40 ml/min a 24 hour urine creatinine clearance can be used.
  * Albumin > 2.5 mg/dL
  * INR ≤ 1.5
* Life expectancy > 6 months
* Capable of giving written informed consent

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen
* Contraindication to receiving radiotherapy
* Prior chemotherapy
* Prior biliary resection or attempted resection
* Prior transperitoneal biopsy
* Large esophageal varices without band ligation
* Active GI bleed or within 2 weeks of study enrollment
* Ascites refractory to medical therapy or shunting
* Active/unresolved biliary tract obstruction
* Presence of multifocal, lymphatic, or extrahepatic metastases
* Participation in another concurrent treatment protocol
* If history of other primary cancer, subject eligible only if she or he has:

  * Curatively resected non-melanomatous skin cancer
  * Curatively treated cervical carcinoma in situ
  * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 3 years
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
* Any psychiatric or other disorder (eg brain metastases) likely to impact on informed consent
* Pregnancy or breast-feeding
* While not excluded, patients with significant impaired hearing must be made aware of potential ototoxicity and may choose not to be included. If included, baseline audiograms are recommended and, in those given cisplatin, should be followed by repeat audiograms prior to cycle 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The location is the Stanford Cancer Center. The study was open to accrual 1/18/2011. The study closed on 9/28/2012.
Groups:
- SBRT, Chemotherapy and Liver Transplantation: The patients received Stereotactic Body Radiotherapy and Chemotherapy followed by a liver transplantation. The chemo could be any combination of the following: Gemcitabine, Cisplatin, Carboplatin, Capecitabine and 5FU
Period: Overall Study
Arm/Group | SBRT, Chemotherapy and Liver Transplantation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SBRT, Chemotherapy and Liver Transplantation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 12 Months
Description: Progression free survival is defined to be the time to progression of disease or death.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- SBRT and Chemo: The patients in this arm receive SBRT and chemo in the hope of surviving long enough to have a liver transplantation
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
participants | 0
Statistical Analysis 1: Comparison: SBRT and Chemo; The median Progression Free Survival (PFS) time as calculated using Kaplan Meier methodology. For PFS both death and progression are counted as events; Test type: Superiority or Other; months = 8.5, 95% CI 2-sided [7 to 10] — There were only two patients in the study. Both died without having any local failure. One patient died at 10 months, the other at 7 months. The range for the 95%CI is both the full range and the 95%CI

2. Secondary Outcome: Pathologic Complete Response Rate
Description: Pathologic complete response will be defined as no residual tumor cells seen on the explanted liver specimen.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
participants | 0

3. Secondary Outcome: Serum CA 19-9 Levels
Description: Initial level of Cancer antigen 19-9
Time Frame: 12 months
Measure: Mean (Full Range); unit: U/ml
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
U/ml | 3329.1 [62.2 to 6596]

4. Secondary Outcome: Overall Survival at 12 Months
Description: the estimated probability for the percentage of participants with overall survival at 12 months.
Time Frame: 12 months
Population: There were only two patients analyzed. Please take that under advisement when looking at the results.
Measure: Number; unit: probability
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
probability | 0

5. Secondary Outcome: Liver Transplant Rate
Description: The number of patients receiving liver transplant among patients who initially have tumors ≤3 cm
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
participants | 0

6. Secondary Outcome: Freedom From Local Progression at 12 Months
Description: the proportion of patients who experienced a local recurrence at 12 months with death as a competing risk
Time Frame: 12 months
Population: Neither of the two patients that participated in the study had a local recurrence prior to dying.
Measure: Number; unit: percentage of patients
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
percentage of patients | 0
Statistical Analysis 1: Comparison: SBRT and Chemo; Test type: Superiority or Other; proportion of participants = 0 — None of the two patients who participated had a local recurrence before they died

7. Secondary Outcome: Liver Transplant Conversion Rate
Description: The ability to successfully perform liver transplant among patients who initially have tumor >3 cm
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
participants | 0

8. Secondary Outcome: Median Time to Overall Survival
Description: The time to overall survival is defined as the time to death from any cause. The median was determined via Kaplan Meier methodology.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT and Chemo
Number analyzed (Participants) | 2
months | 8.5 [7 to 10]

ADVERSE EVENTS:
Time Frame: The entire period of the study, 2 years
Arm/Group | SBRT, Chemotherapy and Liver Transplantation
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT, Chemotherapy and Liver Transplantation (N=2)
Hepatic failure (encephalopathy) (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes